CLINICAL TRIAL: NCT07022652
Title: Influence of Hospital Volume on Mortality and Length of Hospital Stay After Oesophageal Cancer Resection in Switzerland: A Retrospective National Registry Study
Brief Title: Influence of Hospital Volume on Mortality and Length of Hospital Stay After Oesophageal Cancer Resection in Switzerland
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: Hospital volume in ECR
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Esophageal cancer resection — Esophageal cancer resection

SUMMARY:
The effect of centralisation measures on the operative outcomes after oesophageal cancer resection (ECR) in Switzerland has not been highlighted yet. Oesophageal cancer is a rare malignancy in Switzerland. It accounts for 2% of all cancers, with an incidence of 603 per year between 2017 and 2021, affecting primarily men (incidence per year 445, 74%). The mortality of oesophageal cancer is high. The 437 annual oesophageal cancer-related deaths between 2017 and 2021 result in a low 5-year overall survival (OS) of only 30%. Together with the often polymorbid patients, the very demanding surgical technique, and the challenges in postoperative management, a specialised, high-volume, interdisciplinary treatment team is required. The centralisation of such complex surgical procedures in specialised centres aims to build up such treatment teams, resulting in improved quality of the treatment and increased patient safety. To concentrate such procedures in Switzerland, the "Intercantonal agreement on highly specialized medicine" came into force in 2009. In 2013, esophagectomy was regulated for the first time, and the first service allocations were awarded definitely to eight and provisionally to another eight Swiss centres. Before 2013, esophagectomy was performed in 69 hospitals in Switzerland. The decision on the allocation was revised in 2019, resulting in only eight Swiss centres remaining with a service contract for esophagectomy. The next review will take place on the 31st of July 2025.

This retrospective registry study provides Swiss national data on the effect of centralisation on operative outcomes after oesophageal cancer resection (ECR) in Switzerland. It aims to measure the influence of the hospital-specific case number of ECR per year (hospital volume) on the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer resection

Exclusion Criteria:

* Incomplete documentation
* Age under 20 years
* Other hospitals than general or surgical hospitals
* No index operation

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with esophageal cancer resection in Switzerland between 2013 and 2022
Sampling Method: Non-Probability Sample
Enrollment: 2880 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality | Periprocedural
  The association between the hospital volume and the postoperative mortality Mortality Yes or No Hospital volume of esophageal cancer resection as marginal effect Association with GAM logistic regression

SECONDARY OUTCOMES:
Reoperation rate | Periprocedural
  The association between the hospital volume and the reoperation rate Reoperation Yes or No Hospital volume of esophageal cancer resection as marginal effect Association with GAM logistic regression
Length of hospital stay | Periprocedural
  The association between the hospital volume and the length of hospital stay Length of hospital stay in days Hospital volume of esophageal cancer resection as marginal effect Association with quantile regression
Sociodemographic trends | 2013 - 2022

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No